CLINICAL TRIAL: NCT00428753
Title: Matched Case-Control Study of Risk Factors for Human Infection With Avian Influenza A (H5N1) Virus, China
Brief Title: China Case Control Avian Influenza
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0070
Record Dates: First submitted 2007-01-25; First posted 2007-01-30 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Influenza
Keywords: avian influenza, China, H5N1
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

SUMMARY:
This study will determine risk factors of human infection with avian influenza A virus, also known as bird flu virus. Certain risk factors such as exposure to poultry, travel history, health status, and other factors may affect one's risk of getting bird flu. Study participants will include individuals, older than age 1, that tested positive for influenza A (H5N1) in a previous surveillance program and controls (individuals that have not tested positive for avian influenza A (H5N1) and have no fever or respiratory symptoms). There will be 1 study visit during which volunteers will be asked detailed questions about their health, work, and travel habits. Study participants will be asked to donate a blood sample to test for antibodies, the part of the blood that fights infection.

DETAILED DESCRIPTION:
This study is a matched case-control study of risk factors for human infection with avian influenza A (H5N1) virus in China. The primary study objective is to determine the risk factors for avian influenza A (H5N1) virus infection in humans, in China, whether or not the subject was symptomatic. The confirmed case-patients and confirmed antibody positive avian influenza A (H5N1) persons (asymptomatic or sub-clinical) identified by the previously done National Surveillance Program will be included in this study as cases. Controls will be identified from population registries in villages with rural cases and in the adjacent apartment buildings of the urban cases' residences. If the National Surveillance Program identifies healthcare workers infected with avian influenza A (H5N1) virus, healthcare workers in the same department of the healthcare facilities in which the cases worked will also be included as controls. A matched case-control study will be conducted with a ratio of 4 controls per 1 case. Cases and controls who meet the eligibility criteria will be consented and enrolled in the study. After enrollment a questionnaire will be administered to obtain information on demographic characteristics, underlying diseases, daily activities, shopping habits, poultry raising in the backyard, poultry vaccination, exposure to sick/dead poultry or healthy appearing poultry, visits to places where live poultry were kept (e.g., poultry stalls, retail markets, wholesale markets or poultry farms) in the week before illness, eating habits, food preparation activities related to poultry, children's activities such as playing with poultry and swimming in water with water fowl, exposure to other animals including wild birds, and exposure to other humans with respiratory illnesses or confirmed H5N1 case-patients. Survived cases, individuals whose specimen H5N1 tested positive in previous National Surveillance Program and controls will be asked to provide a blood sample to determine whether they have antibodies to H5N1. New confirmed cases and controls will be asked to donate a blood sample for H5N1 antibody testing. Any control that tests positive will become a case and additional controls will be identified. All samples will be tested for H5N1 antibodies with hemagglutination inhibition (using horse red blood cells) and microneutralization assay. If all negative, the individual will be considered sero-negative; if all positive, the individual will be considered sero-positive for the purposes of this study; if results from hemagglutination inhibition (HI) and microneutralization (MN) assays are discordant, the MN result will be considered the final result (negative or positive). Appropriate antigens for the assays will be selected based on the antigenic characteristics of the virus circulating in the region at the time of sample collection. HI and MN assays will be performed according to accepted SOPs. The study will be completed within one year.

ELIGIBILITY:
Inclusion Criteria:

Participants should be informed and assent to participate in this study. For children, informed consent should be provided by their parents or legal guardians. Children aged from 10 years old to 18 years old will be asked to assent.

* Adults or children older than 1 year old.
* Satisfying above definition of cases and controls

Exclusion Criteria:

* Infants younger than 12 months
* For any cases or controls who need proxy, they should be excluded under below situations:

  1. Proxy can not provide sufficient information for this study, or
  2. Proxy refuses to participate in this study, or
  3. No suitable proxy can be found.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2007-01; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Center for Disease Control and Prevention, Beijing, China

REFERENCES:
- [Result] Wang H, Feng Z, Shu Y, Yu H, Zhou L, Zu R, Huai Y, Dong J, Bao C, Wen L, Wang H, Yang P, Zhao W, Dong L, Zhou M, Liao Q, Yang H, Wang M, Lu X, Shi Z, Wang W, Gu L, Zhu F, Li Q, Yin W, Yang W, Li D, Uyeki TM, Wang Y. Probable limited person-to-person transmission of highly pathogenic avian influenza A (H5N1) virus in China. Lancet. 2008 Apr 26;371(9622):1427-34. doi: 10.1016/S0140-6736(08)60493-6. Epub 2008 Apr 8. PMID 18400288